CLINICAL TRIAL: NCT06342102
Title: Pericapsular Nerve Group (PENG) Block and Lateral Femoral Cutaneous Nerve (LFCN) Block Versus Fascia Iliaca (FIC) Block for Multimodal Analgesia After Total Hip Replacement Surgery: a Retrospective Analysis Focused on Movement (Retro- PvF)
Brief Title: PENG and LFCN Block Versus FIC Block for Multimodal Analgesia After Total Hip Replacement Surgery: a Retrospective Analysis Focused on Movement (Retro-PvF)
Acronym: Retro-PvF
Status: Completed | Type: Observational
Sponsor: Ospedale Edoardo Bassini (Other)
Responsible Party: Principal Investigator, Francesco Vetrone, MD, Medical Doctor, Ospedale Edoardo Bassini
Other Study IDs: ID 4286
Record Dates: First submitted 2024-03-26; First posted 2024-04-02 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Regional Anesthesia Block; Regional Anesthesia; Total Hip Replacement Surgery; Total Hip Arthroplasty (THA)
Keywords: PENG; LFCN; fascia iliaca; THA; total hip replacement surgery; analgesia; movement; Peripheral nerve blocks
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- PENG + LFCN Block: group in which PENG + LFCN Block was performed
  Interventions: Procedure: PENG + LFCN block
- FIC Block: group in which FIC Block was performed
  Interventions: Procedure: FIC block

INTERVENTIONS:
Procedure: PENG + LFCN block — The PENG block was performed under ultrasound guidance. After skin disinfection, the needle was advanced between the psoas tendon and pubic ramus where 20 mL of 0.5% ropivacaine were injected. The LFCN block was performed following the PENG block.10 ml of 0.5% ropivacaine were injected near the nerve into the fat-filled flat tunnel (FFFT) located at the level of the superior anterior iliac spine and lateral to the sartorius muscle.
  Other Names: pericapsular nerve group block associated with lateral femoral cutaneous nerve block
  Groups: PENG + LFCN Block
Procedure: FIC block — FICB was performed under ultrasound guidance. The needle was advanced above the fascia iliaca and 20 mL of 0.5% ropivacaine were injected
  Other Names: fascia iliaca compartment block
  Groups: FIC Block

SUMMARY:
Total hip arthroplasty is a major surgical procedure performed on a growing number of patients. Optimal pain control with limited muscle weakness is paramount for a swift initiation of physical therapy and ambulation, thus expediting hospital discharge. Amongst the many peripheral nerve blocks, FIB (fascia iliaca block) has been recommended as the block of choice by many international guidelines since it offers the best pain control with a relatively low risk of motor block. PENG (pericapsular nerve group) and its association with LFCN (lateral femoral cutaneous nerve) has been proposed as an effective alternative that offers comparable, If not better, pain control with a considerably lower risk for motor block compared to FIB. Given the novelty of this block, there are few published papers on the subject, mostly case series or case reports thus justifying the need for retrospective study.

DETAILED DESCRIPTION:
The primary outcome was the degree of residual quadriceps femoris muscle paresis assessed with the MRC (medical research council) scale at 6 hours between PENG and LCFN. The secondary outcomes were NRS (numeric rating scale) at 6,12, 24 hours, total opioid consumption expressed as milligrams of morphine equivalents (MME), time to first rescue opioid and time to first postoperative ambulation.

ELIGIBILITY:
Inclusion Criteria:

* elective total hip replacement surgery for non-traumatic hip disease,
* age over 18 years,
* complete clinical chart including type of peripheral nerve block performed,
* signed consent form for spinal anesthesia and peripheral nerve block.

Exclusion Criteria:

* preoperative opioid therapy,
* having received a peripheral nerve block other than PENG + LFCN or FICB,
* having received general anesthesia,
* incomplete chart,
* documented muscle weakness
* deviation from the established post-operative analgesia protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Historical cohort study conducted among all patients who had THA from November 2022 to October 2023 at the ASST Nord Milano - Bassini Hospital, Cinisello Balsamo, Milano, Italy.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2024-03-26 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Movement of the lower limb affected by surgery | 6 hours after surgery
  The Medical Research Council (MRC) Muscle Strength Scale (ranging scale from 0 to 5 0= no visible contraction, 5=normal power) was used to assess the degree of residual quadriceps femoris muscle paresis 6 hours postoperatively.

SECONDARY OUTCOMES:
pain control | 6 hours after surgery
  pain assessment with Numeric Rating Scale (NRS): a 0-10 scale, with zero meaning "no pain" and 10 meaning "the worst pain imaginable"
pain control | 12 hours after surgery
  pain assessment with Numeric Rating Scale (NRS): a 0-10 scale, with zero meaning "no pain" and 10 meaning "the worst pain imaginable"
pain control | 24 hours after surgery
  pain assessment with Numeric Rating Scale (NRS): a 0-10 scale, with zero meaning "no pain" and 10 meaning "the worst pain imaginable"
Morphine Milligram Equivalents (MME) of "pro re nata" (PRN) opioid doses | 24 hours after surgery
  we studied the effect of Regional anesthesia on opioid-sparing
Morphine Milligram Equivalents (MME) of "pro re nata" (PRN) opioid doses | 6 hours after surgery
  we studied the effect of Regional anesthesia on opioid-sparing
Morphine Milligram Equivalents (MME) of "pro re nata" (PRN) opioid doses | 12 hours after surgery
  we studied the effect of Regional anesthesia on opioid-sparing

OTHER OUTCOMES:
time to first opioid request | From date of surgery until up to 3 days after
  we studied the effect of Regional anesthesia on opioid-sparing
time to first postoperative ambulation | From date of surgery until up to 3 days after
  we studied the effect of Regional anesthesia on opioid-sparing

CONTACTS AND LOCATIONS:
Locations (1):
- ASST Nord Milano - Ospedale E. Bassini, Cinisello Balsamo, Italy/Milano, Italy

IPD SHARING:
Plan to Share IPD: No